CLINICAL TRIAL: NCT00822380
Title: Evaluation of the Efficacy of Different Strategies to Treat Anemia in Mexican Children: A Randomized Clinical Trial
Brief Title: Evaluation of the Efficacy of Different Strategies to Treat Anemia in Mexican Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Dr Jorge Luis Rosado Loria, Universidad Autonoma de Querétaro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNN2002-07
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Anemia
Keywords: Anemia; Iron; Children; Micronutrients
MeSH Terms: conditions — Anemia | interventions — Iron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anemic children (Experimental)
  Interventions: Dietary Supplement: Iron; Dietary Supplement: Multiple micronutrients supplement; Dietary Supplement: micronutrient fortified porridge powder; Dietary Supplement: Iron and ascorbic acid fortified water; Dietary Supplement: Iron plus folic acid supplement

INTERVENTIONS:
Dietary Supplement: Iron — Daily 20mg of ferrous sulfate in liquid solution during 4 months
Dietary Supplement: Multiple micronutrients supplement — Daily supplement with 10mg of iron plus several micronutrients following a formula designed to treat anemia in indigenous population in Mexico. During 4 months.
Dietary Supplement: micronutrient fortified porridge powder — Daily powdered complementary food designed for a national program in Mexico with 10mg of iron plus several micronutrients during 4 months
Dietary Supplement: Iron and ascorbic acid fortified water — A drink water product fortified with 6.7 mg ofiron, zinc and ascorbic acid. This product was asked to be used for drinking and for cooking for the child during 4 months.
Dietary Supplement: Iron plus folic acid supplement — Daily liquid solution following the daily iron (12.5mg)and folic acid recommendation of UNICEF to treat anemia during 4 months

SUMMARY:
Anemia continues to be a major public health problem in many regions of the world and it is still not clear which strategy is more effective in children population in terms of adherence and efficacy. The objective was to evaluate the efficacy and acceptance of several strategies that have been recently recommended to treat anemia on anemic children (6 to 43 mo):Iron supplement, iron+folic acid supplement, a multiple micronutrients supplement a micronutrient fortified complementary food in the form of porridge powder or zinc+iron+ascorbic acid fortified water.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin less than 11.7g/dL and above 7.0g/dL

Exclusion Criteria:

* Breastfeeding
* Chronic gastroenteritis
* Any other severe illness

Ages: 6 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 680 (Actual)
Dates: Start 2003-03; Primary Completion 2003-11 (Actual); Study Completion 2004-11 (Actual)

REFERENCES:
- [Derived] Rosado JL, Gonzalez KE, Caamano Mdel C, Garcia OP, Preciado R, Odio M. Efficacy of different strategies to treat anemia in children: a randomized clinical trial. Nutr J. 2010 Sep 23;9:40. doi: 10.1186/1475-2891-9-40. PMID 20863398